CLINICAL TRIAL: NCT06309225
Title: Pilot Feasibility Trial of Dose Adjusted Chemoradiotherapy in HPV-Associated Oropharynx Cancer of the Elderly (DACHOC-E)
Brief Title: Dose Adjusted Chemoradiotherapy in HPV-Associated Oropharynx Cancer of the Elderly
Acronym: (DACHOC-E)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Omar Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Omar Mahmoud, Principal Investigator, Baptist MD Anderson Cancer Center, Florida
Organization: Baptist MD Anderson Cancer Center, Florida (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMDA-2301
Record Dates: First submitted 2024-02-22; First posted 2024-03-13 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Oropharynx Cancer; Frailty
MeSH Terms: conditions — Oropharyngeal Neoplasms; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Cisplatin: 30-40 mg/m2/week, every week during radiation. Dose should be based on actual body weight. The first cisplatin infusion should be started within 24 hours before or after the first scheduled radiation treatment.
  Intensity Modulated Radiation Therapy (IMRT) and Image-Guided Radiation Therapy (IGRT) are mandatory for this study.
  55 Gy radiation in 5 weeks using 5 fractions per week + Cisplatin every week
  Interventions: Radiation: Modified dose and fields intensity modulated radiotherapy

INTERVENTIONS:
Radiation: Modified dose and fields intensity modulated radiotherapy — Instead of standard bilateral or extensive neck fields, the current radiation fields will cover disease with only 3cm expansion. The clinical target volumes doses are biologically equivalent to the standard but given in a shorter hypofractionated approach.

SUMMARY:
Previous studies of this type of head and necl cancer have shown high rates of cancer control but result in many short and long term side effects when treated with high dose radiation and chemotherapy. Recently, investigators have noticed similar high rates of cancer control in small numbers of patients who receive less intensive treatments using lower doses of radiation, smaller radiation fields with chemotherapy. It is expected that the side effects of treatment with lower doses of radiation would be less.

For this reason this study is looking at a different regimen of reducing the intensity of the treatment.

The purpose of this study is to compare any good and bad effects of using lower dose smaller fields radiation therapy and chemotherapy with published outcomes. This study will allow the researchers to know whether these different approaches are better, the same, or worse than the usual approach. To be better, the study approach should result in the same survival rate of the usual approach (about 85 out of 100 patients alive and free of cancer at 2 years) but with less long-term side effects.

DETAILED DESCRIPTION:
There will be about 30 people taking part in this study. This study has one study group. All the people on the study will receive radiation therapy once a day, 5 days a week (for a total of 55 Gy over 5 weeks) and chemotherapy, cisplatin, (given through the vein for about 30-60 minutes) once a week for 5 weeks.

Medications and saline solutions to prevent side effects of chemotherapy may also be given by vein and may prolong your time in the chemotherapy clinic to as much as 4-6 hours.

Standard regimen not delivered on this study pertains to radiation therapy and chemotherapy, cisplatin in a schedule of 5 treatments a week for a total of 69.96 Gy over 6.5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of squamous cell carcinoma of the oropharynx (tonsil, base of tongue, soft palate, or oropharyngeal walls)
* Patients must have clinically or radiographically evident measurable disease at the primary site or at nodal stations.
* P16-positive based on local site immunohistochemical tissue staining
* Clinical stage T1-3, N1-2, M0 (AJCC, 8th ed.)
* Age ≥ 65.
* Normal organ and marrow function within 14 days prior to registration defined as follows:
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Hemoglobin ≥ 8.0 g/dL
* Total bilirubin ≤ 1.5× institutional upper limit of normal (ULN)
* AST(SGOT) or ALT(SGPT) ≤ 3.0 × institutional ULN
* Serum creatinine ≤ 1.5× ULN

Exclusion Criteria:

* Metastatic disease
* Recurrent disease after primary management Cancers with center of mass is outside the oropharyngeal boundaries
* Synchronous double primaries
* Prior radiotherapy for lymphoma or other malignancy
* Prior systemic therapy including immunotherapy
* Severe active comorbidity where life expectancy is <1 year.
* Autoimmune disease
* Uncontrolled HIV

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Two-year progression free survival | 2 years
  Assuming the primary endpoint (non-inferior 2 year locoregional control) is met and both of these toxicity outcome goals are met, then concurrent short course radiotherapy would be considered an effective and less toxic alternative to concurrent standard arm, in locally advanced HPV-associated carcinoma of the oropharynx.

SECONDARY OUTCOMES:
Benefit and Tolerance of Treatment | 2 years
  Frailty index G8 score 14 as major determinant of benefit and tolerance to treatment through:
  Per prior study score <14 (1-17) is an indicator of frailty. The frailty as a factor in completing therapy (yes or no) and number of days break from therapy will be used as a variable.
  G20 frailty index (G-20 is the actual name and not abbreviation) is as follows:
  A Has food intake declined over the past 3 months due to loss of appetite, digestive problems, chewing or swallowing difficulties? B Weight loss during the last 3 months C Mobility D Neuropsychological problems E Body Mass Index (BMI (weight in kg) / (height in m²) F Takes more than 3 medications per day G In comparison with other people of the same age, how does the patient consider his/her health status? H Age
Acute Toxicity | 2 years
  Acute toxicity (Grade 3 or higher)
Late toxicity | 2 years
  Late toxicity (Grade 3 or higher)
Failure pattern | 2 years
  Pattern failure (local in field, local marginal miss, local regional failure, distant failure, combination of the above).
  As some of the patient may have recurrence in the radiation fields, this will be termed local recurrence. Recurrence outside the radiation fields but in the head and neck area will be quantified as regional failure. Failure outside the head and neck area will be classified as distant failure. This outcome will be quantified as global number of failure out of the 20 patients and their distribution will be quantified in a diagram as explain above.

CONTACTS AND LOCATIONS:
Locations (1):
- Baptist MD Anderson Cancer Center, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-28): https://cdn.clinicaltrials.gov/large-docs/25/NCT06309225/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT06309225/ICF_001.pdf